CLINICAL TRIAL: NCT03572517
Title: Comparison of Two Different Anesthetic Techniques on Incidence of Postoperative Delirium in Cancer Patients After Laparoscopic Surgery in Trendelenburg Position: A Prospective Randomized Clinical Trial
Brief Title: Incidence of Postoperative Delirium in Cancer Patients After Laparoscopic Surgery in Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2205/16
Record Dates: First submitted 2018-02-07; First posted 2018-06-28 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2018-02

CONDITIONS: Delirium; Anesthesia
Keywords: Delirium; Anesthesia; Surgical Oncology
MeSH Terms: conditions — Delirium | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Patients will be allocated sequentially in 2 groups. Sequential allocation will be used in order to control age as a possible confounding factor for the outcome of interest. The randomization will be performed through free software R version 3.4.
  1. Balanced general anesthesia.
  2. Balanced general anesthesia associated with subarachnoid block with 0.5% heavy bupivacaine (3ml).
  All patients will receive morphine 50 mcg via the spinal route.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subarachnoid block (Active Comparator): Subarachnoid block with hyperbaric bupivacaine 0,5% 3ml associate with morphine 50 mcg.
  A general anesthetic with fentanyl 3 mcg / kg + propofol 2 mg / kg + rocuronium 0.6 mg / kg will be performed.
  Anesthesia will be maintained with remifentanil (ng / ml) through Minto's pharmacokinetic model (BBraun infusion syringe - Perfusor® Space model) and desflurane (Fe%).
  Interventions: Procedure: Subarachnoid block
- Spinal morphine (Active Comparator): Spinal morphine with morphine 50 mcg. A general anesthetic with fentanyl 3 mcg / kg + propofol 2 mg / kg + rocuronium 0.6 mg / kg will be performed.
  Anesthesia will be maintained with remifentanil (ng / ml) through Minto's pharmacokinetic model (BBraun infusion syringe - Perfusor® Space model) and desflurane (Fe%).
  Interventions: Procedure: Spinal morphine

INTERVENTIONS:
Procedure: Subarachnoid block — Balanced general anesthesia (Induction of anesthesia: Propofol, fentanyl and rocuronium. Maintenance: Desflurane /remifentanil) associated with subarachnoid block (bupivacaine and morphine)
  Arms: Subarachnoid block
Procedure: Spinal morphine — Balanced general anesthesia (Induction of anesthesia: Propofol, fentanyl and rocuronium. Maintenance: Desflurane /remifentanil) and spinal analgesia with morphine
  Arms: Spinal morphine

SUMMARY:
Postoperative delirium is an acute mental syndrome that is caused by diffuse cerebral dysfunction resulting from the action of predisposing and precipitating factors acting together. It is associated with an increase in mortality and postoperative morbidity and prolongs the period of hospitalization of the patient Videolaparoscopic surgery has been increasingly used as a therapeutic and diagnostic method. In order to have a good visualization of the anatomical structures on which it will act, it is necessary to introduce gas into the cavity, a mandatory component known as pneumoperitoneum. This technique gives special characteristics for the conduction of anesthesia, since the positive intra-abdominal pressure results in changes in the patient's physiology. Some types of laparoscopic surgery require the position of Trendelenburg for better visualization of the operative field. Among the changes related to this position are the increase in cardiac output and intracranial pressure.

In order to optimize the anesthetic procedure, anesthetic blocks have been increasingly used, especially the spinal. The association of general anesthesia with spinal anesthesia, followed by its contraindications is advantageous, because lower doses of anesthetic agents are necessary for the maintenance of general anesthesia. This association results in an earlier awakening, a reduction of nausea / vomiting, postoperative pain, length of hospital stay, cost effectiveness and greater patient satisfaction. As a disadvantage, by associating general anesthesia with spinal anesthesia, patients become susceptible to the adverse events of spinal anesthesia. Among these, the most common are headache, hypotension, nausea and vomiting, pruritus, urinary retention and tremor. Performing spinal anesthesia with opioids alone, without the use of local anesthetic is also possible, with morphine being the most used. The benefit of this variation of technique is analgesia for a period of 12 to 24 hours, without the cardiovascular consequences resulting from the action of the local anesthetic.

JUSTIFICATION: There are no studies in the literature evaluating The objective of this study is to analyze if the anesthetic techniques employed, general anesthesia or general anesthesia associated with subarachnoid block, for videolaparoscopic oncologic surgeries, in Trendelenburg position, differ in relation to the incidence of delirium in the postoperative period.

DETAILED DESCRIPTION:
Patients will be allocated sequentially in 2 groups. Sequential allocation will be used in order to control age as a possible confounding factor for the outcome of interest.

These patients will be monitored intraoperatively with electrocardiogram (ECG), noninvasive pressure, pulse oximetry, capnography, BIS, monitor of neuromuscular blocker (TOF), esophageal temperature and Trendelenburg angle.

The measured moments will be patient entry in the operating room, after pre-anesthetic medication, anesthetic pre-induction, after anesthetic induction, after surgical incision, after pneumoperitoneum infusion, after Trendelenburg position, every 15 minutes until the end of the procedure and after extubation.

All patients will receive morphine 50 mcg via the spinal route. All patients will receive intravenous pre-anesthetic medication midazolam 0.03 mg / kg for comfort during spinal anesthesia and 500 ml of crystalloid solution prior to blockade associated with 4 ml / kg / hour of crystalloid solution plus volume to be depended of clinical parameters.

Subarachnoid block will be performed in the seated position, antisepsis / asepsis with alcoholic chlorhexidine, location of the L3 / L4 space, needle puncture with whitacre 27 G, barbotation of 0.5 ml and injection lasting 5 to 7 seconds.

Spinal morphine will be performed with the same anesthetic technique described in the subarachnoid block.

A general anesthetic with pre-oxygenation 8 liters / minute for 5 minutes + fentanyl 3 mcg / kg + propofol 2 mg / kg + rocuronium 0.6 mg / kg will be performed. Patients will be ventilated with a mixture of oxygen and air through an inspired fraction of 40% oxygen and maintaining an expired concentration of carbon dioxide between 35 and 45 mmHg. Anesthesia will be maintained with remifentanil (ng / ml) through Minto's pharmacokinetic model (BBraun infusion syringe - Perfusor® Space model) and desflurane (Fe%).

Hypnosis will be guided by maintaining BIS between 40 and 60 and the dose of remifentanil will be adjusted by vital signs.

Patients with medium arterial pressure with values lower than 60 mmHg will be medicated with vasopressors depending on heart rate. If heart rate is greater than 60 beats per minute (bpm) metaraminol 0.5 mg will be used and 5 mg ephedrine will be used if heart rate less than 60 bpm.

In both groups, the patients will be kept warm with a thermal blanket and will have their esophageal temperature measured (40 cm from the incisor teeth).

After the surgical procedure, neuromuscular blockade will be antagonized with suggamadex, according to the monitoring of neuromuscular blockade through TOF.

* Deep block (at least 1 to 2 responses in PTC, but prior to the appearance of T2, ie the second response to TOF): 4 mg / kg.
* Moderate block (after onset of T2): 2mg / kg.
* 16 mg / kg is recommended if there is a clinical condition requiring rapid reversal (approximately 3 minutes) following the single dose of rocuronium at 1.2 mg / kg.

After 5 minutes of extubation, vital signs (blood pressure, heart rate, saturation) will be collected and the patient will be evaluated for the presence of delirium. Dipyrone 2 grams and parecoxib 40 mg will be performed without contraindication for postoperative analgesia.

Patients will then be referred to the anesthetic recovery room, where they will continue to be monitored with ECG, noninvasive pressure and pulse oximeters. They will also be evaluated for pain in the numerical estimate scale (NRS) (0 = no pain, up to 10 = maximum pain), on arrival and every 30 minutes until the time of discharge into the room. Those who present pain with NRS greater than 4 in PACU will be treated with morphine 1 mg every 10 minutes. Those with nausea / vomiting will be given alizapride 50 mg.

Patients will be assessed with regard to the appearance of delirium by means of CAM (Confusion Assemption Method) in association with the Richmond Agitation Sedation Scale (RASS) scale.

CAM is a simple screening method based on the following four questions, with Criteria 1 and 2 plus 3 or 4 being present:

1. Acute onset: Is there evidence of acute change in the patient's underlying mental state?
2. Attention Disorder: Has the patient had difficulty focusing on his or her attention, for example, was easily distracted or had difficulty following what was being said?
3. Disorganized thinking: Was the patient's thinking disorganized or incoherent, with dispersive or irrelevant conversion, unclear or illogical flow of ideas, or unpredictable change of subject?
4. Changes in level of consciousness: Does the patient present altered level of consciousness such as lethargy, torporous, comatose? The RASS, was developed with the purpose of characterizing the level of consciousness and agitation. Signs of hyperactive delirium are defined as scores ranging from +1 (anxious patient), +2 (frequent uncoordinated unintentional movements, fight against ventilation), +3 (aggressive) to +4 (very aggressive). Signs of hypoactive delirium are defined as RASS ranging from - 5 (patient does not respond), - 4 (no response to voice sound), -3 (movements or ocular opening to voice sound), -2 (awakens briefly), - 1 (not completely alert) to 0 (patient calm or sleepy).

This evaluation will be performed by nurses, previously trained, on arrival at PACU every 30 minutes until discharge from the post-anesthetic recovery room and 24 hours after the patient's discharge from the hospital. In cases where the patient has an episode of persistent delirium for more than 1 hour, the evaluation of a psychiatrist will be requested for follow-up and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Oncologic patients submitted to elective videolaparoscopic surgery in Trendelenburg position
* 18 years or older
* ASA lesser than 3
* period of at least 2 hours in Trendelenburg position

Exclusion Criteria:

* With absolute contraindication and related to spinal anesthesia
* With difficult airway prediction with possibility of awake intubation.
* With previous diagnosis of: cognitive disorder and / or depression.
* Chronic use of benzodiazepines (use during the last 12 weeks).
* Referred to perform the postoperative ICU.
* With diagnosis of anemia (Hemoglobin <10).
* With diagnosis of current infection.
* With renal disease with stage> G3a (glomerular filtration rate <45 ml / min / 1.73 m2.
* With body mass index (BMI) characterized by obesity (BMI> 30 kg / m2).
* With history of nausea / vomiting in previous anesthetic procedures.
* With diagnosis of malignant hyperthermia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Confusion Assessment Method in association with Richmond Agitation Sedation Scale will be used to postoperative delirium diagnosis. | Until discharge from hospital (an average of 3 days)
  Confusion Assessment Method: presence or absence of delirium
  If present should be classified
  Richmond Agitation Sedation Scale (positive):4 Combative; 3 Very agitated; 2 Agitated;1 Restless 0 Alert and calm (negative):1Drowsy;2 Light sedation; 3 Moderate sedation;4 Deep sedation;5 Unarousable
  (positive) delirium hyperactive (negative) delirium hypoactive

SECONDARY OUTCOMES:
Numeric Pain Rating Scale will be used to evaluate pain. | Until discharge from hospital (an average of 3 days)
  Postoperative pain Number scale from 0 (minimum level of pain) to 10 (higher level of pain)

CONTACTS AND LOCATIONS:
Overall Officials: Giane Nakamura, Study Chair — A.C. Camargo Cancer Center
Locations (1):
- A.C. Camargo Cancer Center, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Absalom AR, Glen JI, Zwart GJ, Schnider TW, Struys MM. Target-Controlled Infusion: A Mature Technology. Anesth Analg. 2016 Jan;122(1):70-8. doi: 10.1213/ANE.0000000000001009. PMID 26516798
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Ali HH, Utting JE, Gray C. Stimulus frequency in the detection of neuromuscular block in humans. Br J Anaesth. 1970 Nov;42(11):967-78. doi: 10.1093/bja/42.11.967. No abstract available. PMID 5488360
- [Background] Ali S, Patel M, Jabeen S, Bailey RK, Patel T, Shahid M, Riley WJ, Arain A. Insight into delirium. Innov Clin Neurosci. 2011 Oct;8(10):25-34. PMID 22132368
- [Background] American Geriatrics Society Expert Panel on Postoperative Delirium in Older Adults. Postoperative delirium in older adults: best practice statement from the American Geriatrics Society. J Am Coll Surg. 2015 Feb;220(2):136-48.e1. doi: 10.1016/j.jamcollsurg.2014.10.019. Epub 2014 Nov 14. No abstract available. PMID 25535170
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Apfel CC, Kranke P, Katz MH, Goepfert C, Papenfuss T, Rauch S, Heineck R, Greim CA, Roewer N. Volatile anaesthetics may be the main cause of early but not delayed postoperative vomiting: a randomized controlled trial of factorial design. Br J Anaesth. 2002 May;88(5):659-68. doi: 10.1093/bja/88.5.659. PMID 12067003
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Araimo Morselli FSM, Zuccarini F, Caporlingua F, Scarpa I, Imperiale C, Caporlingua A, De Biase L, Tordiglione P. Intrathecal Versus Intravenous Morphine in Minimally Invasive Posterior Lumbar Fusion: A Blinded Randomized Comparative Prospective Study. Spine (Phila Pa 1976). 2017 Mar;42(5):281-284. doi: 10.1097/BRS.0000000000001733. PMID 27306255
- [Background] Asfar P, Meziani F, Hamel JF, Grelon F, Megarbane B, Anguel N, Mira JP, Dequin PF, Gergaud S, Weiss N, Legay F, Le Tulzo Y, Conrad M, Robert R, Gonzalez F, Guitton C, Tamion F, Tonnelier JM, Guezennec P, Van Der Linden T, Vieillard-Baron A, Mariotte E, Pradel G, Lesieur O, Ricard JD, Herve F, du Cheyron D, Guerin C, Mercat A, Teboul JL, Radermacher P; SEPSISPAM Investigators. High versus low blood-pressure target in patients with septic shock. N Engl J Med. 2014 Apr 24;370(17):1583-93. doi: 10.1056/NEJMoa1312173. Epub 2014 Mar 18. PMID 24635770
- [Background] Barrio J, Errando CL, San Miguel G, Salas BI, Raga J, Carrion JL, Garcia-Ramon J, Gallego J. Effect of depth of neuromuscular blockade on the abdominal space during pneumoperitoneum establishment in laparoscopic surgery. J Clin Anesth. 2016 Nov;34:197-203. doi: 10.1016/j.jclinane.2016.04.017. Epub 2016 May 11. PMID 27687373
- [Background] Bartels K, Esper SA, Thiele RH. Blood Pressure Monitoring for the Anesthesiologist: A Practical Review. Anesth Analg. 2016 Jun;122(6):1866-79. doi: 10.1213/ANE.0000000000001340. PMID 27195632
- [Background] Bessa SS, Katri KM, Abdel-Salam WN, El-Kayal el-SA, Tawfik TA. Spinal versus general anesthesia for day-case laparoscopic cholecystectomy: a prospective randomized study. J Laparoendosc Adv Surg Tech A. 2012 Jul-Aug;22(6):550-5. doi: 10.1089/lap.2012.0110. Epub 2012 Jun 11. PMID 22686181
- [Background] Birch DW, Dang JT, Switzer NJ, Manouchehri N, Shi X, Hadi G, Karmali S. Heated insufflation with or without humidification for laparoscopic abdominal surgery. Cochrane Database Syst Rev. 2016 Oct 19;10(10):CD007821. doi: 10.1002/14651858.CD007821.pub3. PMID 27760282
- [Background] Borgeat A, Ekatodramis G, Schenker CA. Postoperative nausea and vomiting in regional anesthesia: a review. Anesthesiology. 2003 Feb;98(2):530-47. doi: 10.1097/00000542-200302000-00036. No abstract available. PMID 12552215
- [Background] Brull SJ, Murphy GS. Residual neuromuscular block: lessons unlearned. Part II: methods to reduce the risk of residual weakness. Anesth Analg. 2010 Jul;111(1):129-40. doi: 10.1213/ANE.0b013e3181da8312. Epub 2010 May 4. PMID 20442261
- [Background] Bryson GL. [Methods and madness: agitation, delirium, and postoperative cognitive dysfunction]. Can J Anaesth. 2010 Sep;57(9):799-803. doi: 10.1007/s12630-010-9339-8. No abstract available. French. PMID 20526707
- [Background] Campbell N, Boustani M, Limbil T, Ott C, Fox C, Maidment I, Schubert CC, Munger S, Fick D, Miller D, Gulati R. The cognitive impact of anticholinergics: a clinical review. Clin Interv Aging. 2009;4:225-33. doi: 10.2147/cia.s5358. Epub 2009 Jun 9. PMID 19554093
- [Background] Card E, Pandharipande P, Tomes C, Lee C, Wood J, Nelson D, Graves A, Shintani A, Ely EW, Hughes C. Emergence from general anaesthesia and evolution of delirium signs in the post-anaesthesia care unit. Br J Anaesth. 2015 Sep;115(3):411-7. doi: 10.1093/bja/aeu442. Epub 2014 Dec 23. PMID 25540068
- [Background] Carmichael DE. Laparoscopy-cardiac considerations. Fertil Steril. 1971 Jan;22(1):69-70. doi: 10.1016/s0015-0282(16)37990-0. No abstract available. PMID 5538757
- [Background] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111
- [Background] Closhen D, Treiber AH, Berres M, Sebastiani A, Werner C, Engelhard K, Schramm P. Robotic assisted prostatic surgery in the Trendelenburg position does not impair cerebral oxygenation measured using two different monitors: A clinical observational study. Eur J Anaesthesiol. 2014 Feb;31(2):104-9. doi: 10.1097/EJA.0000000000000000. PMID 24225725
- [Background] Cestari A, Buffi NM, Scapaticci E, Lughezzani G, Salonia A, Briganti A, Rigatti P, Montorsi F, Guazzoni G. Simplifying patient positioning and port placement during robotic-assisted laparoscopic prostatectomy. Eur Urol. 2010 Mar;57(3):530-3. doi: 10.1016/j.eururo.2009.11.028. Epub 2009 Nov 17. PMID 19963314
- [Background] de Boer HD, Driessen JJ, Marcus MA, Kerkkamp H, Heeringa M, Klimek M. Reversal of rocuronium-induced (1.2 mg/kg) profound neuromuscular block by sugammadex: a multicenter, dose-finding and safety study. Anesthesiology. 2007 Aug;107(2):239-44. doi: 10.1097/01.anes.0000270722.95764.37. PMID 17667567
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Fabbri RM, Moreira MA, Garrido R, Almeida OP. Validity and reliability of the Portuguese version of the Confusion Assessment Method (CAM) for the detection of delirium in the elderly. Arq Neuropsiquiatr. 2001 Jun;59(2-A):175-9. doi: 10.1590/s0004-282x2001000200004. PMID 11400020
- [Background] Farag E, Chelune GJ, Schubert A, Mascha EJ. Is depth of anesthesia, as assessed by the Bispectral Index, related to postoperative cognitive dysfunction and recovery? Anesth Analg. 2006 Sep;103(3):633-40. doi: 10.1213/01.ane.0000228870.48028.b5. PMID 16931673
- [Background] Gerges FJ, Kanazi GE, Jabbour-Khoury SI. Anesthesia for laparoscopy: a review. J Clin Anesth. 2006 Feb;18(1):67-78. doi: 10.1016/j.jclinane.2005.01.013. PMID 16517337
- [Background] Golinger RC, Peet T, Tune LE. Association of elevated plasma anticholinergic activity with delirium in surgical patients. Am J Psychiatry. 1987 Sep;144(9):1218-20. doi: 10.1176/ajp.144.9.1218. PMID 3631323
- [Background] Gutt CN, Oniu T, Mehrabi A, Schemmer P, Kashfi A, Kraus T, Buchler MW. Circulatory and respiratory complications of carbon dioxide insufflation. Dig Surg. 2004;21(2):95-105. doi: 10.1159/000077038. Epub 2004 Feb 27. PMID 15010588
- [Background] Henny CP, Hofland J. Laparoscopic surgery: pitfalls due to anesthesia, positioning, and pneumoperitoneum. Surg Endosc. 2005 Sep;19(9):1163-71. doi: 10.1007/s00464-004-2250-z. Epub 2005 Jul 28. PMID 16132330
- [Background] Hirsch J, DePalma G, Tsai TT, Sands LP, Leung JM. Impact of intraoperative hypotension and blood pressure fluctuations on early postoperative delirium after non-cardiac surgery. Br J Anaesth. 2015 Sep;115(3):418-26. doi: 10.1093/bja/aeu458. Epub 2015 Jan 23. PMID 25616677
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Kalmar AF, Foubert L, Hendrickx JF, Mottrie A, Absalom A, Mortier EP, Struys MM. Influence of steep Trendelenburg position and CO(2) pneumoperitoneum on cardiovascular, cerebrovascular, and respiratory homeostasis during robotic prostatectomy. Br J Anaesth. 2010 Apr;104(4):433-9. doi: 10.1093/bja/aeq018. Epub 2010 Feb 18. PMID 20167583
- [Background] Kopman AF, Naguib M. Laparoscopic surgery and muscle relaxants: is deep block helpful? Anesth Analg. 2015 Jan;120(1):51-58. doi: 10.1213/ANE.0000000000000471. PMID 25625254
- [Background] Lepouse C, Lautner CA, Liu L, Gomis P, Leon A. Emergence delirium in adults in the post-anaesthesia care unit. Br J Anaesth. 2006 Jun;96(6):747-53. doi: 10.1093/bja/ael094. Epub 2006 May 2. PMID 16670111
- [Background] Lestar M, Gunnarsson L, Lagerstrand L, Wiklund P, Odeberg-Wernerman S. Hemodynamic perturbations during robot-assisted laparoscopic radical prostatectomy in 45 degrees Trendelenburg position. Anesth Analg. 2011 Nov;113(5):1069-75. doi: 10.1213/ANE.0b013e3182075d1f. Epub 2011 Jan 13. PMID 21233502
- [Background] McDaniel M, Brudney C. Postoperative delirium: etiology and management. Curr Opin Crit Care. 2012 Aug;18(4):372-6. doi: 10.1097/MCC.0b013e3283557211. PMID 22732435
- [Background] Messina AG, Wang M, Ward MJ, Wilker CC, Smith BB, Vezina DP, Pace NL. Anaesthetic interventions for prevention of awareness during surgery. Cochrane Database Syst Rev. 2016 Oct 18;10(10):CD007272. doi: 10.1002/14651858.CD007272.pub2. PMID 27755648
- [Background] O'Malley C, Cunningham AJ. Physiologic changes during laparoscopy. Anesthesiol Clin North Am. 2001 Mar;19(1):1-19. doi: 10.1016/s0889-8537(05)70208-x. PMID 11244911
- [Background] Rex C, Bergner UA, Puhringer FK. Sugammadex: a selective relaxant-binding agent providing rapid reversal. Curr Opin Anaesthesiol. 2010 Aug;23(4):461-5. doi: 10.1097/ACO.0b013e32833a5413. PMID 20489603
- [Background] Rosendal C, Markin S, Hien MD, Motsch J, Roggenbach J. Cardiac and hemodynamic consequences during capnoperitoneum and steep Trendelenburg positioning: lessons learned from robot-assisted laparoscopic prostatectomy. J Clin Anesth. 2014 Aug;26(5):383-9. doi: 10.1016/j.jclinane.2014.01.014. Epub 2014 Jul 30. PMID 25086483
- [Background] Salluh JI, Wang H, Schneider EB, Nagaraja N, Yenokyan G, Damluji A, Serafim RB, Stevens RD. Outcome of delirium in critically ill patients: systematic review and meta-analysis. BMJ. 2015 Jun 3;350:h2538. doi: 10.1136/bmj.h2538. PMID 26041151
- [Background] Sanders RD, Pandharipande PP, Davidson AJ, Ma D, Maze M. Anticipating and managing postoperative delirium and cognitive decline in adults. BMJ. 2011 Jul 20;343:d4331. doi: 10.1136/bmj.d4331. No abstract available. PMID 21775401
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Steiner LA. Postoperative delirium. Part 1: pathophysiology and risk factors. Eur J Anaesthesiol. 2011 Sep;28(9):628-36. doi: 10.1097/EJA.0b013e328349b7f5. PMID 21785356
- [Background] Steiner LA. Postoperative delirium. part 2: detection, prevention and treatment. Eur J Anaesthesiol. 2011 Oct;28(10):723-32. doi: 10.1097/EJA.0b013e328349b7db. PMID 21912241
- [Background] Wang M, Singh A, Qureshi H, Leone A, Mascha EJ, Sessler DI. Optimal Depth for Nasopharyngeal Temperature Probe Positioning. Anesth Analg. 2016 May;122(5):1434-8. doi: 10.1213/ANE.0000000000001213. PMID 26974019
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Wongyingsinn M, Baldini G, Stein B, Charlebois P, Liberman S, Carli F. Spinal analgesia for laparoscopic colonic resection using an enhanced recovery after surgery programme: better analgesia, but no benefits on postoperative recovery: a randomized controlled trial. Br J Anaesth. 2012 May;108(5):850-6. doi: 10.1093/bja/aes028. Epub 2012 Mar 8. PMID 22408272
- [Background] Yu D, Chai W, Sun X, Yao L. Emergence agitation in adults: risk factors in 2,000 patients. Can J Anaesth. 2010 Sep;57(9):843-8. doi: 10.1007/s12630-010-9338-9. Epub 2010 Jun 5. PMID 20526708